CLINICAL TRIAL: NCT01949948
Title: Randomised Trial of Tenecteplase vs. Alteplase for Recanalisation in Acute Ischemic Stroke
Brief Title: Study of Tenecteplase Versus Alteplase for Thrombolysis (Clot Dissolving) in Acute Ischemic Stroke
Acronym: NOR-TEST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lars Thomassen (Other)
Collaborators: The Research Council of Norway (Other)
Responsible Party: Sponsor-Investigator, Lars Thomassen, Senior Consultant neurologist; Professor, Haukeland University Hospital
Organization: Haukeland University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REK 2011/2435
Record Dates: First submitted 2013-09-21; First posted 2013-09-25 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Ischemic Stroke
Keywords: treatment, intervention, thrombolysis
MeSH Terms: conditions — Ischemic Stroke | interventions — Tenecteplase; Tissue Plasminogen Activator

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tenecteplase (Active Comparator): 0.4 mg/kg single bolus intravenously
  Interventions: Drug: Tenecteplase
- Alteplase (Active Comparator): 0.9 mg/kg as 10% bolus + 90% infusion/60 minutes intravenously
  Interventions: Drug: Alteplase

INTERVENTIONS:
Drug: Tenecteplase — 0.4 mg/kg single bolus intravenously
  Other Names: Metalyse
  Arms: Tenecteplase
Drug: Alteplase — 0.9 mg/kg as 10% bolus + 90% infusion/60 minutes intravenously
  Other Names: Actilyse
  Arms: Alteplase

SUMMARY:
BACKGROUND: Alteplase dissolves blood vessel clots in acute ischemic stroke and is the only approved acute drug treatment <4½ hours of stroke onset. The overall benefit from alteplase is substantial, but up to 2/3 of patients with large artery clots may not achieve reopening of the vessel and up to 40% of the patients may remain severely disabled or die, leaving substantial room for improvement. Tenecteplase, widely used in coronary heart disease, may be more effective and may have less bleeding complications than alteplase, and may be the drug of choice also in stroke.

HYPOTHESIS: Tenecteplase may be given safely to patients with acute ischemic stroke at a dose that is associated with improved clinical outcome compared with existing treatment options.

AIMS: To compare efficacy and safety of tenecteplase vs. alteplase given <4½ hours after symptom onset.

STUDY ENDPOINTS: The primary study endpoint is excellent clinical outcome at 3 months (effect). Secondary study endpoints are major early clinical improvement (effect) and bleeding complications (safety).

DETAILED DESCRIPTION:
HYPOTHESIS: 1) Tenecteplase 0.4 mg/kg may be given safely to patients with acute ischaemic stroke <4½ hours after stroke onset. 2) Tenecteplase 0,4 mg/kg (single bolus)has superior efficacy and safety compared with alteplase 0.9 mg/kg (10% bolus + 90% infusion/60 minutes) when given within 4 ½ hours after stroke onset.

DESIGN: NOR-TEST is a multi-centre PROBE (prospective randomised, open-label, blinded endpoint) trial with randomisation tenecteplase:alteplase 1:1.

POWER CALCULATION: NOR-TEST aims at detecting a 9 % higher percentage excellent outcome with tenecteplase vs. alteplase (r1=0.40; r2=0.49; OR 1.44; power 0.8), and will include 954 patients during 3 years.

PATIENT RECRUITMENT: All patients found eligible for thrombolytic therapy are eligible for NOR-TEST, i.e. NOR-TEST changes neither inclusion nor exclusion criteria. The number of patients treated at a participating centre will therefore essentially remain unchanged. Estimated 400 patients are thrombolysed per year in participating centres. Allowing for 20% of patients not being included in NOR-TEST, the total number of patients (n=954) will still be met.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Ischaemic stroke with measurable deficit on NIH Stroke Scale
* All stroke sub-types, severities and vascular distributions,a visible arterial occlusion is not required for inclusion
* Treatment within 4 ½ hours of stroke onset
* Patients awakening with symptoms are defined by the time last observed normal and awake
* Informed written consent signed by the patient, verbal consent from the patients as witnessed by a non-participating health care person, or consent by the signature of the patient's family must be provided

Exclusion Criteria:

* Patients with premorbid modified Rankin Scale (mRS) score ≥3
* Patients for whom a complete NIH Stroke Score cannot be obtained
* Hemiplegic migraine with no arterial occlusion on CTA
* Seizure at stroke onset and no visible occlusion on baseline CTA
* Intracranial haemorrhage on baseline CT
* Clinical presentation suggesting subarachnoid haemorrhage even if baseline CT is normal
* Large areas of hypodense ischaemic changes on baseline CT
* Patients with systolic blood pressure >185 mm Hg or diastolic blood pressure >110 mm Hg
* Female, pregnant or breast feeding
* Known bleeding diathesis
* Use of oral anticoagulants and International Normalized Ratio (INR) ≥1,4
* Use of new oral anticoagulants (NOAC) within the last 12 hours
* Heparin <48 hours and increased Activated partial thromboplastin tike (APTT)
* Low molecular weight heparin(oid) <24 hours
* Any other investigational drug <14 days
* Sepsis
* Patients with arterial puncture at a noncompressible site or lumbar puncture <7 days
* Major surgery or serious trauma <14 days
* Gastrointestinal or urinary tract hemorrhage <14 days
* Clinical stroke <2 months
* History of intracranial haemorrhage
* Brain neurosurgery <2 months
* Serious head trauma <2 months
* Pericarditis
* Any serious medical illness likely to interact with treatment
* Confounding pre-existent neurological or psychiatric disease
* Unlikely to complete follow-up
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1050 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Clinical: Functional handicap | 90 days
  Excellent outcome defined as mRS 0-1

SECONDARY OUTCOMES:
Symptomatic cerebral hemorrhage | 24-36 hours
  Haemorrhagic transformation (haemorrhagic infarct / haematoma) as defined by CT (or MRI)
Hemorrhagic transformation | 24-36 hours
  Any hemorrhagic infarct or parenchymal hematoma
Neurological improvement | 24 hours
  NIHSS changes from baseline: NIHSS=0 or reduction of ≥4 NIHSS points
Clinical: Functional handicap | 90 days
  Ordinal shift analysis of mRS
Safety | 90 days
  Death

CONTACTS AND LOCATIONS:
Overall Officials: Lars Thomassen, MD PhD Prof., Study Chair — Dept. Neurology, Haukeland University HospitalBergen, Norway; Ulrike Waje-Andreassen, MD PhD Prof., Study Director — Dept. Neurology, Haukeland University Hospital, Bergen; Nicola Logallo, MD PhD, Principal Investigator — Dept. Neurology, Haukeland University Hospital, Bergen, Norway
Locations (13):
- Norway (13):
  - Haukeland University Hospital, Bergen
  - Nordland Hospital, Bodø
  - Drammen Hospital, Drammen
  - Førde Central Hospital, Førde
  - Haugesund Hospital, Haugesund
  - Molde Hospital, Molde
  - Akershus University Hospital, Nordbyhagen
  - Ullevål University Hospital, Oslo
  - Baerum Hospital, Rud
  - Telemark Hospital, Skien
  - Stavanger University Hosital, Stavanger
  - St. Olav Hospital NTNU, Trondheim
  - Tønsberg Hospital, Tønsberg

REFERENCES:
- [Background] Logallo N, Kvistad CE, Nacu A, Naess H, Waje-Andreassen U, Asmuss J, Aamodt AH, Lund C, Kurz MW, Ronning OM, Salvesen R, Idicula TT, Thomassen L. The Norwegian tenecteplase stroke trial (NOR-TEST): randomised controlled trial of tenecteplase vs. alteplase in acute ischaemic stroke. BMC Neurol. 2014 May 15;14:106. doi: 10.1186/1471-2377-14-106. PMID 24886064
- [Derived] Ronning OM, Nordby L, Logallo N, Kvistad CE, Kristoffersen ES, Ihle-Hansen H, Ihle-Hansen H, Novotny V, Waje-Andreassen U, Naess H, Thomassen L, Thommessen B. Association between blood pressure and outcome in patients with acute ischemic stroke treated with alteplase. J Stroke Cerebrovasc Dis. 2026 Jan;35(1):108518. doi: 10.1016/j.jstrokecerebrovasdis.2025.108518. Epub 2025 Dec 6. PMID 41360194
- [Derived] Novotny V, Kvistad CE, Naess H, Logallo N, Fromm A, Khanevski AN, Thomassen L. Tenecteplase, 0.4 mg/kg, in Moderate and Severe Acute Ischemic Stroke: A Pooled Analysis of NOR-TEST and NOR-TEST 2A. J Am Heart Assoc. 2023 Oct 17;12(20):e030320. doi: 10.1161/JAHA.123.030320. Epub 2023 Oct 13. PMID 37830342
- [Derived] Ihle-Hansen H, Sandset EC, Ihle-Hansen H, Hagberg G, Thommessen B, Ronning OM, Kvistad CE, Novotny V, Naess H, Waje-Andreassen U, Thomassen L, Logallo N. Sex differences in the Norwegian Tenecteplase Trial (NOR-TEST). Eur J Neurol. 2022 Feb;29(2):609-614. doi: 10.1111/ene.15126. Epub 2021 Oct 4. PMID 34564893
- [Derived] Thommessen B, Naess H, Logallo N, Kvistad CE, Waje-Andreassen U, Ihle-Hansen H, Ihle-Hansen H, Thomassen L, Morten Ronning O. Tenecteplase versus alteplase after acute ischemic stroke at high age. Int J Stroke. 2021 Apr;16(3):295-299. doi: 10.1177/1747493020938306. Epub 2020 Jul 6. PMID 32631157
- [Derived] Ahmed HK, Logallo N, Thomassen L, Novotny V, Mathisen SM, Kurz MW. Clinical outcomes and safety profile of Tenecteplase in wake-up stroke. Acta Neurol Scand. 2020 Nov;142(5):475-479. doi: 10.1111/ane.13296. Epub 2020 Jun 23. PMID 32511749
- [Derived] Kvistad CE, Novotny V, Kurz MW, Ronning OM, Thommessen B, Carlsson M, Waje-Andreassen U, Naess H, Thomassen L, Logallo N. Safety and Outcomes of Tenecteplase in Moderate and Severe Ischemic Stroke. Stroke. 2019 May;50(5):1279-1281. doi: 10.1161/STROKEAHA.119.025041. PMID 31009339
- [Derived] Ronning OM, Logallo N, Thommessen B, Tobro H, Novotny V, Kvistad CE, Aamodt AH, Naess H, Waje-Andreassen U, Thomassen L. Tenecteplase Versus Alteplase Between 3 and 4.5 Hours in Low National Institutes of Health Stroke Scale. Stroke. 2019 Feb;50(2):498-500. doi: 10.1161/STROKEAHA.118.024223. PMID 30602354
- [Derived] Logallo N, Novotny V, Assmus J, Kvistad CE, Alteheld L, Ronning OM, Thommessen B, Amthor KF, Ihle-Hansen H, Kurz M, Tobro H, Kaur K, Stankiewicz M, Carlsson M, Morsund A, Idicula T, Aamodt AH, Lund C, Naess H, Waje-Andreassen U, Thomassen L. Tenecteplase versus alteplase for management of acute ischaemic stroke (NOR-TEST): a phase 3, randomised, open-label, blinded endpoint trial. Lancet Neurol. 2017 Oct;16(10):781-788. doi: 10.1016/S1474-4422(17)30253-3. Epub 2017 Aug 2. PMID 28780236
- [Derived] Logallo N, Kvistad CE, Thomassen L. Therapeutic Potential of Tenecteplase in the Management of Acute Ischemic Stroke. CNS Drugs. 2015;29(10):811-8. doi: 10.1007/s40263-015-0280-9. PMID 26387127